CLINICAL TRIAL: NCT02526264
Title: Clinical Trial to Evaluate Quality of Life, Period of Hospitalization and Complication Rates in Patients With Stoma Receiving Specific Preoperative Education vs. Standard Preoperative Education
Brief Title: Evaluation of Quality of Life and Period of Hospitalization by Education
Acronym: STELLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STELLA
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
Keywords: stoma; quality of life
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Krankenhaus Nordwest Concept (Experimental): specific preoperative education program realised by a specialized stoma-therapist containing individualized information on material maintenance, hygiene, nutrition, complications, activities of daily life and occupation
  Interventions: Other: Education program
- Standard concept (Experimental): standard preoperative education program administered by a surgeon containing information on surgery, outcome, risks and alternatives
  Interventions: Other: Education program

INTERVENTIONS:
Other: Education program — Verbal education prior tu surgery administered to all patients in order to inform about the surgery and outcomes

SUMMARY:
Patients with colorectal cancer prior to stoma surgery are randomized to different preoperative education programs: (a) specific preoperative education, (b) standard preoperative education. Outcome measures are quality of life, period of hospitalization and complication rates.

DETAILED DESCRIPTION:
The present study is initiated to evaluate quality of life, period of hospitalization and complication rates in patients with colorectal cancer receiving treatment with stoma surgery. Prior to surgery patients are randomized to different preoperative education programs. In Arm A patients receive a new specific education program (Krankenhaus Nordwest concept) conducted by a specialized therapist (stoma-therapist). In Arm B patients receive the standard preoperative education program. Standardized questionnaires are used to evaluate quality of life and period of hospitalization at baseline and four weeks after surgery in Arm A vs. Arm B

ELIGIBILITY:
Inclusion Criteria:

* Planned stoma
* colorectal cancer, from resection of left hemi-colon aboral A. colica media
* Patients speaking german and living in Germany
* ECOG ≤ 3
* Informed Consent
* standard education program

Exclusion Criteria:

* Patients treated with stoma by emergency
* patients with dementia
* status post stoma
* Patients in contact with a stoma-therapist
* recurrence of colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2015-11-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 9-15 days after surgery
  Quality of life is assessed with EORTC QLQ-30 and EORTC QLQ-CR 29 at baseline, 9-15 days after surgery and 4 weeks after surgery. An improvement in Arm A is characterized by 10 points
Quality of Life | 4 weeks after surgery
  Quality of life is assessed with EORTC QLQ-30 and EORTC QLQ-CR 29 at baseline, 9-15 days after surgery and 4 weeks after surgery. An improvement in Arm A is characterized by 10 points

SECONDARY OUTCOMES:
Period of hospitalization | 9-15 days after surgery, 4 weeks after surgery
Complication rates | 9-15 days after surgery, 4 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Krankenhaus Nordwest, Frankfurt
  - Sana Klinikum, Offenbach

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared